CLINICAL TRIAL: NCT01842984
Title: Increasing Social Competence and Social Integration of Older Adults Experiencing Loneliness
Brief Title: Decreasing Loneliness in Older Adults
Acronym: I-SOCIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Ministry for Senior Citizens, Israel (Unknown)
Responsible Party: Principal Investigator, Professor Jiska Cohen-Mansfield, Professor, Department of Health Promotion, Director- The Minerva Center for the Interdisciplinary Study of the End of Life, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300009673
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Loneliness; Social Isolation
Keywords: Loneliness; Social isolation; Depression; Older adults; Social competence; Social integration
MeSH Terms: conditions — Social Isolation; Depression; Social Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-SOCIAL intervention (Experimental): Participants in this group will have up to 10 personal meetings with activities counselors and several group meetings.
  Interventions: Behavioral: I-SOCIAL intervention
- Control group (No Intervention): Participants in this group will not have meetings with the activities counselors, and will not take part in the group meetings.

INTERVENTIONS:
Behavioral: I-SOCIAL intervention — The I-SOCIAL intervention is based on findings from Cohen-Mansfield and Parpura-Gill (2007), which highlighted the important role of barriers in contributing to loneliness in older persons. These barriers include a perceived lack of opportunities for social contacts, low social self-efficacy, and health and mobility difficulties. The intervention includes: (1) identifying the barriers for the specific person; (2) up to 10 meetings with an activities counselor. The meetings include discussions concerning options for social contacts and use of techniques and resources to tackle the barriers; and (3) group meetings of participants and the activities counselors in order to provide a concrete social event and as a venue to discuss barriers and ways to address them.
  Arms: I-SOCIAL intervention

SUMMARY:
The purposes of this study are: (1) decrease loneliness and social isolation and increase social competence and social integration of older adults experiencing loneliness; (2) examine an intervention process grounded in a theoretical model that was developed in a previous study. The intervention process is tailored to the participants' barriers and abilities, and includes up to 10 personal meetings with an activities counselor and several group meetings.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or over
* residing in the Tel Aviv region

Exclusion Criteria:

* having known mental illness including schizophrenia, depression, bipolar disorder, and dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Loneliness | Participants will be assessed before and after the intervention, an expected average of 6 months
  Loneliness will be assessed via several measures: (a) Frequency of loneliness will be measured via one item ("How often would you say you feel lonely?"; (Mullins, Woodland, & Putnam, 1990) on a 6-point scale from "never" (1) to "several times an hour" (6); (b) The UCLA Loneliness Scale- 8 items (ULS-8; (Hays & DiMatteo, 1987). Each item is rated on a 5-point scale from "not at all" (1) to "to a great extent" (5), with a higher score indicating more loneliness. Based on experience from another study (Cohen-Mansfield et al., 2013) one item ("I am unhappy being so withdrawn") was replaced with two items ("I feel physically distant from other people"; "I feel emotionally distant from other people).

CONTACTS AND LOCATIONS:
Overall Officials: Jiska Cohen-Mansfiels, Professor, Principal Investigator — Tel Aviv University
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided